CLINICAL TRIAL: NCT02156336
Title: A Double-Blind, Placebo-Controlled, Randomized, Parallel Assignment, U.S. Study of Ranolazine for the Treatment of Patients With Diabetic Peripheral Neuropathic Pain (DPNP)
Brief Title: Ranolazine for Diabetic Peripheral Neuropathic Pain (DPNP)
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Not enough patients met study criteria for enrollment.
Sponsor: Horizons International Peripheral Group (Other)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HIPG-CLIN-2014-01
Record Dates: First submitted 2014-05-28; First posted 2014-06-05 (Estimated); Last update posted 2017-02-10 (Actual); Status verified 2017-02

CONDITIONS: Diabetic Peripheral Neuropathic Pain
Keywords: Diabetic Peripheral Neuropathic Pain; Ranexa; Ranolazine; Neurology
MeSH Terms: interventions — Ranolazine; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- PLACEBO (Placebo Comparator): * 500 mg PLACEBO PO 2 times a day for 1 week (Week 1)
  * 1000 mg PLACEBO PO 2 times a day for 5 weeks (Weeks 2,3,4,5,6)
  Interventions: Drug: Placebo
- RANOLAZINE (Active Comparator): * 500 mg RANOLAZINE PO 2 times a day for 1 week (Week 1)
  * 1000 mg RANOLAZINE PO 2 times a day for 5 weeks (Weeks 2,3,4,5,6)
  Interventions: Drug: Ranolazine

INTERVENTIONS:
Drug: Ranolazine — Oral administration, BID; for a maximum of 51 days.
  Other Names: Ranexa
  Arms: RANOLAZINE
Drug: Placebo — Oral administration, BID; for a maximum of 51 days.
  Other Names: Sugar Pill
  Arms: PLACEBO

SUMMARY:
The purpose of this trial is to determine if patients suffering from diabetic peripheral neuropathic pain treated with ranolazine will have a greater reduction in pain compared to placebo.

Hypothesis: From the prior clinical observations, and analgesic efficacy in the preclinical animal model of neuropathic pain, the investigators hypothesize that subjects randomized to ranolazine will show a greater reduction in diabetic neuropathic pain compared to placebo.

ELIGIBILITY:
Inclusion Criteria:

1. A minimum of 18 years of age;
2. Provided signed Informed Consent Form and Health Insurance Portability and Accountability Act (HIPAA) authorization for this study approved by the Institutional Review Board;
3. Patients must have diabetic peripheral neuropathic pain rated at an average level of six (6) or above as documented in daily diary prior to baseline visit and noted at Baseline Visit;
4. Diabetic on a stable insulin regimen or oral medication regimen as determined by the investigator [It is recommended Hba1c < 9.5%, making a note that lab normal values may vary among sites.];
5. Clinical Exam Results:

   1. 5.07 Semmes-Weinstein Monofilament Test Subject does not sense monofilament or evokes an abnormal response in a minimum of two (2) out of five (5) test locations on the plantar surface of the foot.
   2. Pin Prick Test Subject experiences allodynia, hyperalgesia, or sensory loss in two (2) out of five (5) test locations in the plantar surface - four (4) and dorsum - one (1) of the foot.
6. Willing and able to comply with the requirements of the protocol and follow directions from the clinic and research staff;
7. For female patients only:

   * Be post-menopausal (no menses for at least 2 years) or sterilized,
   * If subject of childbearing potential, not breastfeeding, has a negative pregnancy test at Baseline (pre-randomization, Day 0), has no intention of becoming pregnant during the course of the study, and is using one or more of the following contraceptive measures:

     1. Stable regimen of hormonal contraception
     2. Intra-uterine device
     3. Condoms with spermicide
     4. Diaphragm with spermicide

Exclusion Criteria:

1. History of allergy or intolerance to ranolazine;
2. Any condition or concomitant medication that would preclude the safe use of ranolazine as outlined in the prescribing information sheet;
3. In the judgment of the investigator, any clinically-significant ongoing medical condition that might jeopardize the patient's safety or interfere with the absorption, distribution, metabolism or excretion of the study drug;
4. In the judgment of the investigator, clinically-significant abnormal physical findings during screening (excluding the patient's peripheral neuropathy condition);
5. Use participation in another experimental or investigational drug or device trial;
6. Pregnant or breast feeding;
7. Cirrhosis of the liver;
8. Psychological or addictive disorders (not limited to, but including for example, drug and/or alcohol dependency) that may preclude patient consent or compliance, or that may confound study interpretation;
9. Taking a moderate or strong CYP3A inhibitor (e.g. diltiazem, verapamil, ketoconazole, itraconazole, clarithromycin, erythromycin, nefazodone, nelfinavir, ritonavir, indinavir, and saquinavir);
10. Taking inducers of Cytochrome P450, family 3, subfamily A (CYP3A) (e.g. rifampin, rifabutin, rifapentine, phenobarbital, phenytoin, carbamazepine, and St. John's wort);
11. Renal impairment as defined by a calculated serum creatinine clearance of < 30ml/min;
12. Lower back disorders where symptoms present similarly to DPNP;
13. Family history of long QT syndrome;
14. Congenital long QT syndrome;
15. Subjects taking tricyclic antidepressants;
16. Subjects taking anti-psychotic drugs;
17. Patient is taking > 850mg metformin BID;
18. Any subjects currently taking pregabalin;
19. Any subjects currently taking gabapentin;
20. Any subject currently taking Metanx®;
21. Any subjects currently taking continuous long-term narcotics;
22. Grapefruit and grapefruit containing products;
23. Use of P-gp inhibitors - cyclosporine.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2014-05; Primary Completion 2017-02-08 (Actual); Study Completion 2017-02-08 (Actual)

PRIMARY OUTCOMES:
Fifty percent or greater reduction in the mean Numeric Rating Scale (11-point NRS 0-10) recorded in the subjects' diaries from ranolazine compared to placebo. | 6 weeks (42 Days)

SECONDARY OUTCOMES:
Change in Quality of Life Assessment as measured by SF-36 v2 | Randomization (Day 0) and Day 42
Change in pain assessment measured by the Visual Analog Scale | Randomization (Day 0), Day 14, Day 28, Day 42, and Day 56
Change in pain assessment measured by Short-Form McGill Pain Questionnaire | Randomization (Day 0) and Day 42
Change in pain of patients with arterial ischemia measured by Short-Form McGill Pain Questionnaire | Randomization (Day 0), Day 14, Day 28, Day 42, and Day 56
  Pain reduction of ranolazine versus placebo in subjects with diabetic peripheral neuropathic pain (DPNP) and arterial ischemia compared to those with DPNP without arterial ischemia.
Additional pain medication | Randomization (Day 0), Day 14, Day 28, Day 42, and Day 56
  Additional pain medication after the baseline visit as needed for pain reduction in addition to the study drug.
Occurrence of Adverse Events after randomization | 56 Days
  The rates and severity of Adverse Events (AEs) from Randomization (Day 0) through Termination (Day 56)
Occurrence of Serious Adverse Events after randomization | 56 Days
  A serious adverse event (SAE), also may be called a serious adverse drug reaction, is any untoward medical occurrence that at any dose:
  * results in death,
  * is life-threatening,
  * requires inpatient hospitalization or prolongation of existing hospitalization,
  * results in persistent or significant disability/incapacity, or
  * is a congenital anomaly/birth defect.

CONTACTS AND LOCATIONS:
Overall Officials: Craig M Walker, MD FACC, Principal Investigator — Cardiovascular Institute of the South
Locations (3):
- United States (3):
  - Cardiology Associates, Fairhope, Alabama
  - Cardiovascular Institute of the South, Houma, Louisiana
  - Cardiovascular Institute of the South, Lafayette, Louisiana

REFERENCES:
- [Background] Gould HJ 3rd, Garrett C, Donahue RR, Paul D, Diamond I, Taylor BK. Ranolazine attenuates behavioral signs of neuropathic pain. Behav Pharmacol. 2009 Dec;20(8):755-8. doi: 10.1097/FBP.0b013e3283323c90. PMID 19773645